CLINICAL TRIAL: NCT04129827
Title: Retrospective Cohort Study on How Meniscal Lesions Affect Return to Sport After Anterior Cruciate Ligament Reconstruction in Young Non-professional Athletes
Brief Title: Meniscal Lesions in Return to Sport After Anterior Cruciate Ligament Reconstruction
Acronym: LCA-40
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Collaborators: Istituto di Fisiologia Clinica CNR (Other)
Responsible Party: Principal Investigator, Biagio Moretti, MD, Full Professor, University of Bari
Other Study IDs: 5836
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: ACL Injury; Meniscus Lesion; Sport Injury
Keywords: Return to Sport; ACL reconstruction; Knee; Athletes
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical, self-reported psychological and biomechanical assessments — 1. medical check up
     * active and passive Range Of Motion (ROM)
     * anterior drawer test
     * knee's alignment
     * modified cincinnati rating system questionnaire (mCRSQ)
     * tegner lysholm knee scoring scale (TLKS)
     * Tegner Activity Level Score (TALS)
  2. self-reported psychological questionnaires
     * Tampa Scale of Kinesiophobia (TSK)
     * ACL Return to Sport after Injury (ACL-RSI) score
  3. biomechanical tests
     * Stability test: to balance on one/two legs on a free to move disc for 30s
     * Jump test: i) a maximize jump with both legs; ii) a maximize jump with only one leg; three consecutive jumps; iv) jump coordination path where the patient had to perform a forward-backward-forward jump and a sideway jump on one leg
     * Coordination test: a square hurdle was used for the quick test, where the patient had to step in and out with both feet for a total of 15-rep as quickly as possible
     * fatigue test: to rise and sit from a chair for 30-rep as quickly and safely as possible
  Other Names: CLIMB Battery

SUMMARY:
Most athletes who undergo Anterior Cruciate Ligament Reconstruction (ACLR) plan to return to some level of sporting (RTS) activity. However, rates of return to pre-injury sport are often less than might be expected and many factors influence whether individuals return to sport after this surgery. This study aims to better understand the role of meniscal lesions in RTS and to assess the advantage of the integrated evaluation with clinical, biomechanical and psychological tests to decide the correct RTS timing in non-professional athletes undergoing ACLR.

DETAILED DESCRIPTION:
Twenty non-professional athletes with acute ACL injury were recruited in the Orthopaedic and Trauma Unit of University Hospital of Bari. All the patients underwent an all-inside semitendinosus (ST) tendon autograft ACLR with Arthrex TightRope cortical fixation.

The clinical outcomes (modified Cincinnati Rating System Questionnaire (mCRSQ), Tegner Activity Level Score (TALS), Tegner Lysholm Knee Scoring Scale (TLKSS)), the self-reported psychological scores (Tampa Scale of Kinesiophobia (TSK) and the ACL Return to Sport after Injury (ACL-RSI) score) and biomechanical outcomes (stability, jump, coordination and fatigue tests) were assessed postoperatively at 18 months.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-35 years old
* non professional athletes
* ACLR between January 2017 and December 2017
* all-inside semitendinosus (ST) tendon autograft ACLR with Arthrex TightRope cortical fixation

Exclusion Criteria:

* diabetes
* BMI > 30 kg/m2
* heart disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the patients has been enrolled according to the eligible criteria in Orthopaedic and Trauma Unit of University Hospital of Bari
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between TSK, ACL-RSI Score and mCRSQ Score | 18-months
  Tampa Scale of Kinesiophobia is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.
  ACL Return to Sport after Injury measures the patient's understanding of his knee. It comprises 12 questions with a score of 1 to 10 for each. It is considered that for a normal population without knee condition, the score is between 80 and 90%.
  modified Cincinnati Rating System Questionnaire has been designed to give your therapist information as to how your knee pain has affected your ability to manage in everyday life. It consists of 12 questions, 8 of which are included in the summary score. The total score is calculated as the sum of all questions responses, with 100 representing the best/excellent knee function, and 0 representing the worst/poor knee function.
Correlation between clinical and psychological features | 18-months
  Clinical assessment consist of three tests carried on during medical check-up: i) active and passive Range Of Motion (ROM); ii) anterior drawer test; iii) knee's alignment. All these measurements will be transformed in categorical variables in order to perform chi square test.
Association between clinical features and level of stability | 18-months
  Clinical assessment consist of three tests carried on during medical check-up: i) active and passive Range Of Motion (ROM); ii) anterior drawer test; iii) knee's alignment. All these measurements will be transformed in categorical variables.
  During the stability test, the patient stands with one and two legs respectively on a free to move balance disc for 30 seconds. Subjects were instructed to stand in the centre with their arms at their sides. Level of stability is defined as an index ranking from 1 (low stability) to 5 (high stability).
  Eta square between categorical variables from clinical assessment and the measure outcomes of biomechanical assessment will be performed.
Association between clinical features and limb symmetry index | 18-months
  Clinical assessment consist of three tests carried on during medical check-up: i) active and passive Range Of Motion (ROM); ii) anterior drawer test; iii) knee's alignment. All these measurements will be transformed in categorical variables.
  During jump tests, the subject carried a belt around their hips, and the sensor was placed above the greater trochanter of the hip. Before jumping, the subject had to stand in an upright and still position. A sequence of four different jumps has been executed. The limb symmetry index (LSI) was calculated by dividing the measured value of the injured leg by the value of the non-affected side and multiplying by 100.
  Eta square between categorical variables from clinical assessment and the time required to perform the test will be calculated.
Association between clinical features and Coordination Time | 18-months
  Clinical assessment consist of three tests carried on during medical check-up: i) active and passive Range Of Motion (ROM); ii) anterior drawer test; iii) knee's alignment. All these measurements will be transformed in categorical variables.
  The subject performed one-footed jumps through the course of red (forward-backward-forward jumps) and blue (sideway jumps) hurdles, completing 16 jumps. This had to be performed as quickly as possible by jumping on one leg without a rest between the hurdles.
  Eta square between categorical variables from clinical assessment and the time required to perform the test will be calculated.

SECONDARY OUTCOMES:
Odds ratio between presence of ML and CLIMB-based criteria | 18-months
  The CLIMB battery is the combination of biomechanical, clinical and psychological criteria which could allow to return to sport with the lowest possible risk of reinjury. After performing a correlation matrix and calculating collinearity using linear regression, we will calculate odds ratio as measure of association for presence-absence of meniscal lesion in the observed cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Moretti, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Locations (1):
- Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, IT, Italy

REFERENCES:
- [Result] Bortone I, Moretti L, Bizzoca D, Caringella N, Delmedico M, Piazzolla A, Moretti B. The importance of biomechanical assessment after Return to Play in athletes with ACL-Reconstruction. Gait Posture. 2021 Jul;88:240-246. doi: 10.1016/j.gaitpost.2021.06.005. Epub 2021 Jun 8. PMID 34126566